CLINICAL TRIAL: NCT05569941
Title: A Phase 1, Blinded, Placebo-Controlled Study of the Safety, Tolerability, Pharmacokinetics of Single and Multiple Ascending Doses of ABI-4334 in Healthy Subjects
Brief Title: A First in Human Study to Assess Safety, Tolerability, Pharmacokinetics of ABI-4334 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assembly Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABI-4334-101
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Chronic Hepatitis B
Keywords: ABI-4334; PK; Healthy Subjects
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Part A: SAD Cohorts 1-5 ABI-4334 Tablet (Experimental): A single dose of ABI-4334 will be administered on Day 1 in dose-escalation cohorts with a starting dose of 30 mg. The doses for subsequent cohorts will be determined by evaluation of safety and PK data from previous cohorts.
  Interventions: Drug: ABI-4334 Tablet
- Part A: SAD Cohorts 1-5 ABI-4334 Placebo Tablet (Placebo Comparator): A single dose of placebo matching ABI-4334 will be administered on Day 1.
  Interventions: Drug: ABI-4334 Placebo
- Part A: SAD Fed Cohorts 6-7 ABI-4334 Tablet (Experimental): A single dose of ABI-4334 will be administered after a high-fat meal on Day 1 in cohort 6. A single dose of ABI-4334 will be administered on two separate occasions, once fasted and once after a high-fat meal in cohort 7. The dose administered will be determined after evaluation of cumulative safety and PK data from cohorts 1-5.
  Interventions: Drug: ABI-4334 Tablet
- Part A: SAD Fed Cohorts 6 ABI-4334 Placebo Tablet (Placebo Comparator): A single dose of placebo matching ABI-4334 will be administered on Day 1 after a high-fat meal on Day 1 in cohort 6.
  Interventions: Drug: ABI-4334 Placebo
- Part B: MAD Cohorts 1-2 ABI-4334 Tablet (Experimental): Once-daily doses of ABI-4334 will be administered from Day 1 to Day 8. Cohort B1 will receive a dose determined from evaluation of the data from the SAD cohorts. The doses for the subsequent cohort will be determined by evaluation of safety and PK data from previous cohorts.
  Interventions: Drug: ABI-4334 Tablet
- Part B: MAD Cohorts 1-2 ABI-4334 Placebo Tablet (Placebo Comparator): Once-daily doses of placebo matching ABI-4334 will be administered from Day 1 to Day 8.
  Interventions: Drug: ABI-4334 Placebo

INTERVENTIONS:
Drug: ABI-4334 Tablet — ABI-4334 Tablet
  Arms: Part A: SAD Cohorts 1-5 ABI-4334 Tablet; Part A: SAD Fed Cohorts 6-7 ABI-4334 Tablet; Part B: MAD Cohorts 1-2 ABI-4334 Tablet
Drug: ABI-4334 Placebo — Placebo to ABI-4334 Tablet
  Arms: Part A: SAD Cohorts 1-5 ABI-4334 Placebo Tablet; Part A: SAD Fed Cohorts 6 ABI-4334 Placebo Tablet; Part B: MAD Cohorts 1-2 ABI-4334 Placebo Tablet

SUMMARY:
This study is designed to assess safety, tolerability, and PK of single ascending doses (SAD) of ABI-4334 in Part A and multiple-ascending doses (MAD) of ABI-4334 in Part B in healthy subjects. Effect of food will also be evaluated in Part A.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.0 and 30.0 kg/m2
* In good health (as determined by the Investigator) based on medical history, physical examination, ECG, and clinical laboratory results.
* Female subjects must be non-pregnant and have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Day 1
* Agreement to comply with protocol-specified contraceptive requirements

Exclusion Criteria:

* Positive results for any of the following serology tests, HBsAg, hepatitis B core antibody (HBcAb IgM), hepatitis C virus antibody (HCV Ab), or HIV-1 or -2 antibody
* History of any illness that, in the opinion of the Investigator, might confound the results of the study, pose an additional risk in administering study drug to the subject, or a condition known to interfere with the absorption/ distribution/elimination of drugs.
* History of any significant drug-related allergic reactions such as anaphylaxis, Stevens-Johnson syndrome, urticaria, or multiple drug allergies
* History of persistent alcohol abuse or illicit drug abuse within 3 years prior to Screening
* Has participated in a clinical study involving administration of either an investigational or a marketed drug within 2 months before Screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with adverse events (AEs), premature treatment discontinuation due to AEs, and abnormal laboratory results | Up to Day 14

SECONDARY OUTCOMES:
SAD Cohorts 1-7: Area Under the Plasma Concentration Time Curve (AUC) of ABI-4334 | before and at pre-specified time points up to 144 hours after dosing
SAD Cohorts 1-7: Maximum Observed Plasma Concentration (Cmax) of ABI-4334 | before and at pre-specified time points up to 144 hours after dosing
SAD Cohorts 1-7: Time to Cmax (Tmax) of ABI-4334 | before and at pre-specified time points up to 144 hours after dosing
SAD Cohorts 1-7: Apparent Terminal Elimination Half Life (t 1/2) of ABI-4334 | before and at pre-specified time points up to 144 hours after dosing
SAD Cohorts 1-7: Apparent Systemic Clearance (CL/F) of ABI-4334 | before and at pre-specified time points up to 144 hours after dosing
SAD Cohorts 1-7: Apparent Volume of Distribution (Vz/F) of ABI-4334 | before and at pre-specified time points up to 144 hours after dosing
SAD Cohorts 1-7: Comparison of Cmax between fasted and fed treatments of ABI-4334 | before and at pre-specified time points up to 144 hours after dosing
SAD Cohorts 1-7: Comparison of AUC between fasted and fed treatments of ABI-4334 | before and at pre-specified time points up to 144 hours after dosing
MAD Cohorts 1-2: AUC of ABI-4334 | before and at pre-specified time points up to 24 hours after dosing on Day 1; before dosing on days 2-7; before and up to 120 hours after dosing on Day 8
MAD Cohorts 1-2: Cmax of ABI-4334 | before and at pre-specified time points up to 24 hours after dosing on Day 1; before dosing on days 2-7; before and up to 120 hours after dosing on Day 8
MAD Cohorts 1-2: Tmax of ABI-4334 | before and at pre-specified time points up to 24 hours after dosing on Day 1; before dosing on days 2-7; before and up to 120 hours after dosing on Day 8
MAD Cohorts 1-2: t 1/2 of ABI-4334 | before and at pre-specified time points up to 24 hours after dosing on Day 1; before dosing on days 2-7; before and up to 120 hours after dosing on Day 8
MAD Cohorts 1-2: CL/F of ABI-4334 | before and at pre-specified time points up to 24 hours after dosing on Day 1; before dosing on days 2-7; before and up to 120 hours after dosing on Day 8
MAD Cohorts 1-2: Vz/F of ABI-4334 | before and at pre-specified time points up to 24 hours after dosing on Day 1; before dosing on days 2-7; before and up to 120 hours after dosing on Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Edward Gane, Principal Investigator — New Zealand Clinical Research
Locations (1):
- New Zealand Clinical Research, Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/41/NCT05569941/Prot_SAP_000.pdf